CLINICAL TRIAL: NCT04918147
Title: Elotuzumab in Immunoglobulin G4-Related Disease (IgG4-RD)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated early based on disease flare/lack of efficacy in the early phase of the trial.
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Autoimmunity Centers of Excellence (Other); Bristol-Myers Squibb (Industry); Rho Federal Systems Division, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: DAIT AIG01; UM1AI144298 (NIH); NIAID CRMS ID#: 38708 (Other: DAIT NIAID)
Record Dates: First submitted 2021-06-04; First posted 2021-06-08 (Actual); Results first posted 2025-02-25 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: IgG4 Related Disease; IgG4-RD
Keywords: immune-mediated fibroinflammatory disease; prospective trial; safety and efficacy; IgG4-RD Responder Index (IgG4-RD RI)
MeSH Terms: conditions — Immunoglobulin G4-Related Disease | interventions — elotuzumab; Saline Solution; Methylprednisolone; Methylprednisolone Hemisuccinate; Diphenhydramine; Acetaminophen; Famotidine; Histamine H2 Antagonists; Prednisone; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1a: Elotuzumab-One-Month Regimen (Open-Label) + Pred Taper (Experimental): Per protocol: Six participants will receive elotuzumab on days 0,7, 14, 21, and the prescribed 10-week prednisone taper.
  * Elotuzumab: 10 mg/kg administered once weekly, intravenously for 4 doses, per protocol.
  * Prednisone taper (Pred Taper): Prescribed 10-week dosing taper beginning on Day 0 (baseline) that is taken orally (by mouth) daily, per protocol. Dosage in milligrams (mgs).
  Interventions: Drug: elotuzumab; Drug: methylprednisolone; Drug: diphenhydramine; Drug: acetaminophen; Drug: famotidine; Drug: prednisone
- Cohort 1b: Elotuzumab-Twelve-Month Regimen (Open-Label) + Pred Taper (Experimental): Per protocol: Six participants will receive elotuzumab over a 48 week period, dose of 10mg/kg IV x 1, at baseline, then at weeks 8, 16, 24, 32 and 40 (for a total of 6 doses), with the prescribed 10-week prednisone taper.
  * Elotuzumab: 10 mg/kg administered as referenced above, intravenously, per protocol.
  * Prednisone taper (Pred Taper): Prescribed 10-week dosing taper beginning on Day 0 (baseline) that is taken orally (by mouth) daily, per protocol. Dosage in milligrams (mgs).
  Interventions: Drug: elotuzumab; Drug: methylprednisolone; Drug: diphenhydramine; Drug: acetaminophen; Drug: famotidine; Drug: prednisone
- Cohort 2: Arm A- Elotuzumab (Randomized) + Pred Taper (Experimental): Safety and efficacy analyses from Cohort 1a and Cohort 1b will occur prior to initiating Cohort 2 (Randomized).
  Assuming no safety signal for Cohort 1, forty-two participants will receive elotuzumab per the regimen prescribed above in Part 1B, with the prescribed 10-week prednisone taper.
  * Elotuzumab: 10 mg/kg administered as referenced above, intravenously, per protocol.
  * Prednisone taper (Pred Taper): Prescribed 10-week dosing taper beginning on Day 0 that is taken daily by mouth, per protocol. Dosage in milligrams (mgs).
  Interventions: Drug: elotuzumab; Drug: methylprednisolone; Drug: diphenhydramine; Drug: acetaminophen; Drug: famotidine; Drug: prednisone
- Cohort 2: Arm B-Placebo (Randomized) + Pred Taper (Placebo Comparator): Safety and efficacy analyses from Cohort 1a and Cohort 1b will occur prior to initiating Cohort 2 (Randomized).
  Twenty-one participants will receive placebo for elotuzumab on day 0, then weeks 8, 16, 24, 32 and 40, and the prescribed 10-week prednisone taper.
  * Placebo for elotuzumab: Administered on same schedule as elotuzumab described in Cohort 2 Arm A: intravenously, per protocol.
  * Prednisone taper (Pred Taper): Prescribed 10-week dosing taper beginning on Day 0 taken daily by mouth, per protocol. Dosage in milligrams (mgs).
  Interventions: Drug: placebo for elotuzumab; Drug: methylprednisolone; Drug: diphenhydramine; Drug: acetaminophen; Drug: famotidine; Drug: prednisone

INTERVENTIONS:
Drug: elotuzumab — Elotuzumab is a humanized recombinant monoclonal antibody (mAb) targeted against SLAMF7, a cell surface glycoprotein.
  Other Names: BMS-901608; Empliciti®
  Arms: Cohort 1a: Elotuzumab-One-Month Regimen (Open-Label) + Pred Taper; Cohort 1b: Elotuzumab-Twelve-Month Regimen (Open-Label) + Pred Taper; Cohort 2: Arm A- Elotuzumab (Randomized) + Pred Taper
Drug: placebo for elotuzumab — The placebo for elotuzumab is 0.9% sterile normal saline for injection.
  Other Names: normal saline
  Arms: Cohort 2: Arm B-Placebo (Randomized) + Pred Taper
Drug: methylprednisolone — Premedication administered intravenously, 45 to 90 minutes prior to each elotuzumab/placebo infusion, per protocol. Dosage in milligrams (mg).
  Other Names: Solu-Medrol®
Drug: diphenhydramine — Premedication administered orally or intravenously, 45 to 90 minutes prior to each elotuzumab/placebo infusion, per protocol. Dosage in milligrams (mg).
  Other Names: Benadryl®
Drug: acetaminophen — Premedication administered orally, 45 to 90 minutes prior to each elotuzumab/placebo infusion, per protocol. Dosage in milligrams (mg).
  Other Names: Tylenol®
Drug: famotidine — Premedication administered orally or intravenously, 45 to 90 minutes prior to each elotuzumab/placebo infusion, per protocol. Dosage in milligrams (mg).
  Other Names: H2 blocker
Drug: prednisone — Prescribed dosing with prednisone begins on the day of the first elotuzumab/placebo infusion, administered orally. The ten-week dosing taper proceeds, per protocol. Dosage in milligrams (mg).
  Other Names: corticosteroid

SUMMARY:
This is a two-part multi-center clinical trial in participants with active IgG4-RD.

Part 1 (Cohort 1a and Cohort 1B) is an open-label, dose escalation phase to determine the safety of elotuzumab for investigation in IgG4-RD.

Part 2 (Cohort 2) is a randomized, placebo-controlled, double-blinded (masked) trial phase to compare the effects of elotuzumab and prednisone to elotuzumab placebo and prednisone in participants with IgG4 RD.

Approximately 75 participants with active IgG4-RD will be enrolled in the overall program, 12 in Part 1 and 63 in Part 2. Randomization in Part 2: 2 to 1, with approximately forty-two participants randomized to elotuzumab plus prednisone taper, and twenty-one participants randomized to placebo for elotuzumab plus prednisone taper.

The total duration of participation for each participant in this trial will be 48 weeks (11 months).

DETAILED DESCRIPTION:
Immunoglobulin G4-Related Disease (IgG4-RD) is a chronic fibro-inflammatory condition that can affect virtually every organ system, including the pancreas, biliary tract, salivary and lacrimal glands, orbits, lungs, kidneys, meninges, pituitary gland, prostate and thyroid. It may also involve the retroperitoneum. This multi-organ immune-mediated condition, once regarded as a group of isolated, single-organ diseases, is now recognized to be an overarching, single-disease entity linked by common histopathological and immunohistochemical features.

IgG4-RD tends to afflict middle-aged to elderly individuals. Although IgG4-RD can affect a single organ at presentation, it is not uncommon for participants to present with or develop multi-organ disease. As the disease progresses, additional organs develop lesions and the cellular inflammation characterizing early disease moves toward a more fibrotic stage, causing major tissue damage, dysfunction and ultimately organ failure. It is unclear whether IgG4 itself is involved in the pathogenesis of the disease.

The goals of IgG4-RD treatment are to reduce inflammation and organ swelling and to prevent or reverse tissue fibrosis. No approved therapy exists for IgG4-RD.

This study will enroll adult participants who meet the 2019 American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) Classification Criteria for IgG4-RD, and who have active IgG4-RD with disease manifestations in at least two organ systems.

Primary study objectives:

* To determine the safety and tolerability of the addition of elotuzumab to prednisone in participants with IgG4-RD, and
* To compare the effect of the addition of elotuzumab versus placebo to prednisone on the IgG4-RD Responder Index (IgG4-RD RI), a measure of IgG4-RD disease activity.

ELIGIBILITY:
Inclusion Criteria:

Individuals who meet all of the following criteria are eligible for enrollment as study participants:

1. Participant must be able to understand and provide informed consent and be willing to comply with study procedures and follow up.
2. Are at least 18 years of age and not older than 70 years of age at screening.
3. Meet the ACR/EULAR Classification Criteria for IgG4-RD [30, 31].
4. Have active disease based at screening on an IgG4-RD RI ≥4, with disease manifestations in at least two organ systems.
5. May have newly-diagnosed or relapsing disease at screening. Relapsing disease is defined as IgG4-RD that has previously been in remission but is now active again.
6. May be on treatment or off treatment for IgG4-RD at the time of screening. If on treatment, must be willing to discontinue those other treatments before the baseline visit.
7. No history of severe allergic reactions to monoclonal antibodies.
8. Female participants of childbearing potential must have a negative pregnancy test upon study entry.
9. Female participants of childbearing potential and male participants with a partner of childbearing potential must agree to consistently and correctly use FDA approved highly effective methods of birth control for the entire duration of the study and 6 months after last elotuzumab infusion.
10. Immunization with one of the FDA authorized or licensed SARS-CoV-2 vaccines as per CDC recommendations at the time of informed consent is required for study entry. Vaccinations must have been completed at least 2 weeks prior to start of study therapy.

Exclusion Criteria:

Individuals who meet any of these criteria are not eligible for enrollment as study participants:

1. Presence of a condition other than IgG4-RD that (e.g., asthma) is likely to require systemic Glucocorticoids (GC) for disease control during the period of the trial.
2. Malignancy within 5 years (except successfully treated in situ cervical cancer, resected squamous cell or basal cell carcinoma of the skin.)
3. The following lab values as indicators of hepatic dysfunction:

   1. Serum aspartate aminotransferase (AST) or alanine aminotransferase (ALT) greater than three times the upper limit of normal (ULN)
   2. Total bilirubin > two times the ULN unless caused by Gilbert's disease. Gilbert's disease with total bilirubin > three times ULN.
   3. Serum albumin < 2.5 gm/dL.
4. Evidence of another uncontrolled condition which, in the judgment of the investigator, could interfere with participation in the trial according to the protocol.
5. Active infection requiring hospitalization or treatment with systemic antimicrobial agents within the 30 days prior to treatment allocation/randomization.
6. Prior use of rituximab or other B cell depleting agents within 9 months of enrollment unless B cells have been demonstrated to have repopulated.
7. Use of any investigational agent or biologic and non-biologic DMARDs within 5 half-lives of the agent (or 6 months if the half-life is unknown) prior to enrollment.
8. Any of the following laboratory tests at the Screening Visit:

   1. White blood cell count (WBC) < 3.0 x 103/µL.
   2. Absolute neutrophil count (ANC) < 1.5 x 103/µL.
   3. Hemoglobin < 10 g/dL.
   4. Platelet count < 75 x 109/L.
   5. Estimated glomerular filtration rate (eGFR) ≤ 45 ml/minute/1.73 m2.
9. The use of supplemental oxygen at baseline.
10. At or within 90 days of screening: Positive Interferon-Gamma Release Assay (IGRA). Indeterminate IGRAs must be repeated (with same or other IGRA per local policy) and shown to be negative. Alternatively, if the assay remains indeterminant, a participant must have a negative PPD. Finally, if the participant has had the Bacille Calmette-Guerin (BCG) vaccine or has some other condition complicating the interpretation of TB testing, consultation with infectious disease specialist must be obtained before receipt of the first investigational infusion.

    a. Participants diagnosed with latent TB are eligible but must have received appropriate prophylaxis for 30 days before their first investigational infusion.
11. Medical history or serologic evidence at Screening of chronic infections including:

    1. Human immunodeficiency virus infection.
    2. Hepatitis B as indicated by surface antigen or hepatitis B core antibody positivity
    3. Hepatitis C as indicated by anti-hepatitis C antibody positivity; if a participant is Hepatitis C antibody positive, they will be eligible to participate in the study if he/she is negative for viral load at Screening.
12. Live vaccines within 8 weeks of initiating study therapy.
13. Participant is pregnant or breastfeeding, or planning a pregnancy while enrolled in the study.
14. Substance use disorder, including the recurrent use of alcohol and/or drugs within the past year associated with clinically significant impairment associated with failure to meet major responsibilities at work, school, or home.
15. IgG4-RD that is dominated primarily by advanced fibrotic lesions. Specifically, participants whose disease manifestations consist only of

    1. retroperitoneal fibrosis,
    2. fibrosing mediatinitis,
    3. sclerosing mesenteritis, or
    4. Riedel's thyroiditis. Participants with these disease manifestations can be included, however, only if they have disease in 2 organ systems that is not of an advanced fibrotic nature and otherwise meet the Inclusion and Exclusion Criteria.
16. Evidence a SARS-CoV-2 (COVID-19) infection started within the 30 days prior to treatment allocation/randomization. Participants diagnosed with SARS-CoV-2 (COVID-19) infection more than 30 days prior to treatment allocation/randomization must have symptoms resolved and be deemed fit to participate in the trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-10-13 (Actual); Primary Completion 2024-01-04 (Actual); Study Completion 2024-01-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John H. Stone, MD, MPH, Study Chair — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Emory Healthcare, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic: Pulmonary and Critical Care Medicine, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: Yes
The plan is to share data upon completion of the study in: Immunology Database and Analysis Portal (ImmPort), a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.
Time Frame: On average, within 24 months after database lock for the trial.
Access Criteria: Open access.
URL: https://www.immport.org/home

REFERENCES:
- [Background] Wallace ZS, Naden RP, Chari S, Choi HK, Della-Torre E, Dicaire JF, Hart PA, Inoue D, Kawano M, Khosroshahi A, Lanzillotta M, Okazaki K, Perugino CA, Sharma A, Saeki T, Schleinitz N, Takahashi N, Umehara H, Zen Y, Stone JH; Members of the ACR/EULAR IgG4-RD Classification Criteria Working Group. The 2019 American College of Rheumatology/European League Against Rheumatism classification criteria for IgG4-related disease. Ann Rheum Dis. 2020 Jan;79(1):77-87. doi: 10.1136/annrheumdis-2019-216561. Epub 2019 Dec 3. PMID 31796497
- [Background] Khosroshahi A, Wallace ZS, Crowe JL, Akamizu T, Azumi A, Carruthers MN, Chari ST, Della-Torre E, Frulloni L, Goto H, Hart PA, Kamisawa T, Kawa S, Kawano M, Kim MH, Kodama Y, Kubota K, Lerch MM, Lohr M, Masaki Y, Matsui S, Mimori T, Nakamura S, Nakazawa T, Ohara H, Okazaki K, Ryu JH, Saeki T, Schleinitz N, Shimatsu A, Shimosegawa T, Takahashi H, Takahira M, Tanaka A, Topazian M, Umehara H, Webster GJ, Witzig TE, Yamamoto M, Zhang W, Chiba T, Stone JH; Second International Symposium on IgG4-Related Disease. International Consensus Guidance Statement on the Management and Treatment of IgG4-Related Disease. Arthritis Rheumatol. 2015 Jul;67(7):1688-99. doi: 10.1002/art.39132. No abstract available. PMID 25809420
- See also: Autoimmunity Centers of Excellence (ACE) — https://www.autoimmunitycenters.org/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Three study sites were activated in the United States, beginning in October 2021. A total of nine participants were screened from October 2021 to October 2023 at two sites. Six participants were enrolled in Cohort 1a. Two participants were enrolled in Cohort 1b; enrollment in Cohort 1b was terminated early No participants were enrolled in Part 2.
Groups:
- Cohort 1a: Elotuzumab, 1-Month Regimen + Prednisone Taper: Elotuzumab was administered open label as an intravenous infusion, 10 mg/kg (based on participant's actual weight), on Days 0, 7, 14, 21. Pre-medication with methylprednisolone, diphenhydramine, acetominophen, and an H2 blocker (famotidine or equivalent) occurred prior to each elotuzumab infusion. Participants also received a standardized prednisone taper, starting at either 40 mg orally daily or 30 mg orally based on doses received during the screening period. This was tapered to discontinuation over a 10-week period.
- Cohort 1b: Elotuzumab, 12-Month Regimen + Prednisone Taper: Elotuzumab was administered open label as an intravenous infusion, 10 mg/kg (based on participant's actual weight), on Day 0 and Weeks 8, 16, 24, 32, and 40. Pre-medication with methylprednisolone, diphenhydramine, acetominophen, and an H2 blocker (famotidine or equivalent) occurred prior to each elotuzumab infusion. Participants also received a standardized prednisone taper, starting at either 40 mg orally daily or 30 mg orally based on doses received during the screening period. This was tapered to discontinuation over a 10-week period.
Period: Overall Study
Arm/Group | Cohort 1a: Elotuzumab, 1-Month Regimen + Prednisone Taper | Cohort 1b: Elotuzumab, 12-Month Regimen + Prednisone Taper
Started | 6 | 2
Completed | 6 | 0
Not Completed | 0 | 2
Not completed — Disease flare as defined in protocol | 0 | 2

BASELINE CHARACTERISTICS:
Population: Enrolled
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1a: Elotuzumab, 1-Month Regimen + Prednisone Taper | Cohort 1b: Elotuzumab, 12-Month Regimen + Prednisone Taper | Total
Number analyzed (Participants) | 6 | 2 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 4 | 0 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.8 (6.27) | 56.0 (0.00) | 61.9 (6.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 5 | 0 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 2 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 5 | 0 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 2 | 8
IgG4-Related Disease Responder Index (IgG4-RD RI) Total Activity Score [Mean (Standard Deviation); unit: Scores on a scale] — The IgG4-RD RI detects changes in disease activity for more than 25 organs/sites. It records the following for each: (i) activity trend (through a 0-3 [normal/resolved - worsening]; (ii) presence of symptoms due to active disease; (iii) need for urgent care; (iv) presence of damage; (v) presence of symptoms due to damage. Total activity score is obtained by summing all organ/site activity scores (i) and doubling items needing urgent care (iii). activity scores range from 0 (no active disease) to more than 156 (highest disease activity). Higher scores represent greater (worse) disease activity.
  Scores on a scale | 9.3 (3.01) | 7.0 (4.24) | 8.8 (3.20)

OUTCOME MEASURES:

1. Primary Outcome: The Percent of Participants in Each Cohort Who Experience at Least One Grade 3 or Higher Adverse Event (AE).
Description: The severity of AEs were classified using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE), version 5.0
Time Frame: Up to Week 48 post treatment initiation
Population: The safety population includes all participants who received any amount of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1a: Elotuzumab, 1-Month Regimen + Prednisone Taper | Cohort 1b: Elotuzumab, 12-Month Regimen + Prednisone Taper
Number analyzed (Participants) | 6 | 2
Participants | 5 | 1

2. Secondary Outcome: The Percent of Participants Who Experience at Least One Grade 2 or Higher Adverse Event (AE).
Description: The severity of AEs was classified using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE), version 5.0.
Time Frame: Up to Week 48 post treatment initiation
Population: The safety population includes all participants who received any amount of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1a: Elotuzumab, 1-Month Regimen + Prednisone Taper | Cohort 1b: Elotuzumab, 12-Month Regimen + Prednisone Taper
Number analyzed (Participants) | 6 | 2
Participants | 6 | 2

3. Secondary Outcome: The Percent of Participants With a Grade 3 or Higher Infection
Description: The number of AEs classified as infections that were Grade 3 or higher. The severity of AEs was classified using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE), version 5.0.
Time Frame: Up to Week 48 post treatment initiation
Population: The safety population includes all participants who received any amount of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1a: Elotuzumab, 1-Month Regimen + Prednisone Taper | Cohort 1b: Elotuzumab, 12-Month Regimen + Prednisone Taper
Number analyzed (Participants) | 6 | 2
Participants | 3 | 0

4. Secondary Outcome: The Percent of Participants Who Experience a Malignancy.
Description: The number of participants with malignancies reported as AEs. The severity of AEs was classified using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE), version 5.0.
Time Frame: Up to Week 48 post treatment initiation
Population: The safety population includes all participants who received any amount of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1a: Elotuzumab, 1-Month Regimen + Prednisone Taper | Cohort 1b: Elotuzumab, 12-Month Regimen + Prednisone Taper
Number analyzed (Participants) | 6 | 2
Participants | 0 | 0

5. Secondary Outcome: The Percent of Participants Who Experience a Hepatotoxicity
Description: Hepatotoxicity is defined as an increase in the aspartate aminotransferase (AST) or alanine aminotransferase (ALT) to elevations three times the upper limit of normal.
Time Frame: Up to Week 48 post treatment initiation
Population: The safety population includes all participants who received any amount of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1a: Elotuzumab, 1-Month Regimen + Prednisone Taper | Cohort 1b: Elotuzumab, 12-Month Regimen + Prednisone Taper
Number analyzed (Participants) | 6 | 2
Participants | 0 | 0

6. Secondary Outcome: The Percent of Participants Who Experience a Serious Adverse Event
Description: An adverse event (AE) is considered "serious" if, in the view of either the investigator or sponsor, it results in any of the following outcomes (21 CFR 312.32(a)):
  1. Death. 2. Life-threatening event: An AE is considered "life-threatening" if, in the view of either the investigator or Sponsor, its occurrence places the participant at immediate risk of death. It does not include an AE that, had it occurred in a more severe form, might have caused death. 3. Inpatient hospitalization or prolongation of existing hospitalization. 4. Persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions. 5. Congenital anomaly or birth defect. 6. Important medical events that may not result in death, be life threatening, or require hospitalization may be considered serious when, based upon appropriate medical judgment, they may jeopardize the participant and may require medical or surgical intervention to prevent one of the outcomes listed above.
Time Frame: Up to Week 48 post treatment initiation
Population: The safety population includes all participants who received any amount of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1a: Elotuzumab, 1-Month Regimen + Prednisone Taper | Cohort 1b: Elotuzumab, 12-Month Regimen + Prednisone Taper
Number analyzed (Participants) | 6 | 2
Participants | 4 | 0

7. Secondary Outcome: The Percent of Participants Who Experience Infusion Reactions
Description: The number of participants with infusion reactions reported as AEs. Infusion reactions are defined as any adverse reaction within 24 hours of infusion which are Grade 2 or higher events and at least possibly related to study drug. The severity of AEs was classified using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE), version 5.0.
Time Frame: Up to 24 hours post treatment infusion
Population: The safety population includes all participants who received any amount of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1a: Elotuzumab, 1-Month Regimen + Prednisone Taper | Cohort 1b: Elotuzumab, 12-Month Regimen + Prednisone Taper
Number analyzed (Participants) | 6 | 2
Participants | 1 | 0

8. Secondary Outcome: The Percent of Participants That Reach the Following Threshold Levels of IgG4-Related Disease Responder Index (IgG4-RD RI) Improvement at 24 Weeks: 50% and 75%.
Description: The IgG4-RD RI detects change in disease activity and identifies improvements/worsening in the same or different organ systems. It encompasses more than 25 organs/sites and records the following for each organ/site: (i) activity trend (through a 0-3 [normal/resolved - worsening] organ/site score); (ii) presence of symptoms due to active disease; (iii) need for urgent care; (iv) presence of damage; and (v) presence of symptoms due to damage. The final activity score at each visit is obtained by summing all organ/site scores (i) and by doubling items needing urgent care (iii). Higher scores represent greater (i.e. worse) disease activity. % improvement in the IgG4-RD RI = 100 x ( (Baseline IgG4-RD RI Activity Score - Week 24 IgG4-RD RI Activity Score) / Baseline IgG4-RD RI Activity Score). Participants who use glucocorticoids/immunosuppressants beyond that permitted by protocol, or who experience a disease flare before 24 weeks will be defined as achieving no disease response (0%).
Time Frame: Baseline and Week 24
Population: The safety population includes all participants who received any amount of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1a: Elotuzumab, 1-Month Regimen + Prednisone Taper | Cohort 1b: Elotuzumab, 12-Month Regimen + Prednisone Taper
Number analyzed (Participants) | 6 | 2
Participants
  50% Improvement | 2 | 0
  75% Improvement | 2 | 0

9. Secondary Outcome: Number of Participants With Disease Flares
Description: IgG4-Related Disease flare was defined as recurrence of disease activity such that additional immunosuppressive therapy beyond the trial protocol is indicated. Such additional therapy may include glucocorticoids or alternative immunosuppressive agents. At the time of a potential disease flare, investigators documented the features of the disease flare in each involved organ, including laboratory evaluations, radiology studies, and other procedures (e.g., biopsy). Disease flares were reported as adverse events.
Time Frame: Up to Week 48 post treatment initiation
Population: The safety population includes all participants who received any amount of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1a: Elotuzumab, 1-Month Regimen + Prednisone Taper | Cohort 1b: Elotuzumab, 12-Month Regimen + Prednisone Taper
Number analyzed (Participants) | 6 | 2
Participants | 4 | 2

10. Secondary Outcome: Change From Baseline in Physician Global Assessment
Description: The Physician Global Assessment of the participant's current disease activity was recorded on a 100 mm linear horizontal visual analog scale, where the left hand extreme of the line is considered "Very Good" (0 mm, symptom free and no IgG4-RD symptoms) and the right hand extreme is considered "Very Bad" (100 mm, maximum IgG4-RD activity). Only active disease (as opposed to damage) is considered in the scoring. Change was calculated as the value at Week 12, 24 or 48 minus the value at Baseline.
Time Frame: Baseline, Weeks 12, 24 and 48
Population: The safety population includes all participants who received any amount of investigational product.
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | Cohort 1a: Elotuzumab, 1-Month Regimen + Prednisone Taper | Cohort 1b: Elotuzumab, 12-Month Regimen + Prednisone Taper
Number analyzed (Participants) | 6 | 2
millimeter
  Week 12: number analyzed (Participants) | 0 | 2
  Week 12 |  | 3.0 (24.04)
  Week 24: number analyzed (Participants) | 6 | 0
  Week 24 | -18.5 (15.60) |
  Week 48: number analyzed (Participants) | 6 | 0
  Week 48 | -30.0 (17.32) |

11. Secondary Outcome: Change From Baseline in Patient Global Assessment
Description: The Patient Global Assessment of the participant's current disease activity was recorded on a 100 mm linear horizontal visual analog scale, where the left hand extreme of the line is considered "Very Good" (0 mm, symptom free and no IgG4-RD symptoms) and the right hand extreme is considered "Very Bad" (100 mm, maximum IgG4-RD activity). Change was calculated as the value at Week 12, 24 or 48 minus the value at Baseline.
Time Frame: Baseline, Weeks 12, 24 and 48
Population: The safety population includes all participants who received any amount of investigational product.
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | Cohort 1a: Elotuzumab, 1-Month Regimen + Prednisone Taper | Cohort 1b: Elotuzumab, 12-Month Regimen + Prednisone Taper
Number analyzed (Participants) | 6 | 2
millimeter
  Week 12: number analyzed (Participants) | 0 | 2
  Week 12 |  | -15.0 (32.53)
  Week 24: number analyzed (Participants) | 6 | 0
  Week 24 | 18.8 (40.53) |
  Week 48: number analyzed (Participants) | 6 | 0
  Week 48 | 17.0 (34.04) |

12. Secondary Outcome: Disease-Related Damage, as Measured by the Damage Section of the IgG4-Related Disease (IgG4-RD) Responder Index.
Description: An assessment of damage caused by IgG4-RD in each affected organ is part of the Responder Index. The IgG4-RD RI encompasses more than 25 organs/sites and records the following set of information for each organ/site: (i) activity trend (through a 0-3 [normal/resolved - worsening] organ/site score); (ii) presence of symptoms due to active disease; (iii) need for urgent care; (iv) presence of damage; and (v) presence of symptoms due to damage. Activity and damage are considered separately from the standpoint of scoring, because only disease activity can be expected to respond to treatment. Damage is defined as organ dysfunction that has occurred as a result of IgG4-RD and is considered permanent. The total damage score at each visit is defined as the total number of damaged organs and can range from 0 (no damage) to more than 26 (severe damage).
Time Frame: Screening and Week 24
Population: The safety population includes all participants who received any amount of investigational product.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Cohort 1a: Elotuzumab, 1-Month Regimen + Prednisone Taper | Cohort 1b: Elotuzumab, 12-Month Regimen + Prednisone Taper
Number analyzed (Participants) | 6 | 2
Scores on a scale
  Screening | 1.3 (1.21) | 0 (0)
  Week 24: number analyzed (Participants) | 6 | 0
  Week 24 | 1.5 (1.52) |

ADVERSE EVENTS:
Time Frame: Up to Week 48 post treatment initiation.
Arm/Group | Cohort 1a: Elotuzumab, 1-Month Regimen + Prednisone Taper | Cohort 1b: Elotuzumab, 12-Month Regimen + Prednisone Taper
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/2
Serious Adverse Events (participants affected / at risk) | 4/6 | 0/2
Other Adverse Events (participants affected / at risk) | 6/6 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1a: Elotuzumab, 1-Month Regimen + Prednisone Taper (N=6) | Cohort 1b: Elotuzumab, 12-Month Regimen + Prednisone Taper (N=2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1a: Elotuzumab, 1-Month Regimen + Prednisone Taper (N=6) | Cohort 1b: Elotuzumab, 12-Month Regimen + Prednisone Taper (N=2)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cushing's syndrome (Endocrine disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Immunoglobulin G4 related disease (Immune system disorders) | 4 (4) | 2 (2)
Secondary immunodeficiency (Immune system disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood albumin decreased (Investigations) | 1 (1) | 0 (0)
Blood potassium increased (Investigations) | 1 (1) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Bone cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Failure to achieve remission along with risk of organ damage with disease flare observed in the Cohort 1b participants led to the conservative decision to stop the trial. Last Cohort 1b visit completed was Week 16; no participants enrolled in Part 2.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-19): https://cdn.clinicaltrials.gov/large-docs/47/NCT04918147/Prot_SAP_002.pdf
  • Informed Consent Form (2023-05-19): https://cdn.clinicaltrials.gov/large-docs/47/NCT04918147/ICF_001.pdf